CLINICAL TRIAL: NCT02655510
Title: An Open-Label, Cohort Dose Escalation Study to Assess the Safety and Efficacy of F-652 in Patients With Alcoholic Hepatitis
Brief Title: Use of F-652 in Patients With Alcoholic Hepatitis
Acronym: TREAT 008
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Indiana University (Other); Virginia Commonwealth University (Other); Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Principal Investigator, Vijay Shah, M.D., PI, Mayo Clinic
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-003249
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — eflepedocokin alfa

STUDY DESIGN:
Intervention Model Description: A phase 2 dose escalating study was carried out. F-652 (10, 30 or 45 μg/kg) administered on day 1 and 7 was tested in 3 patients each with moderate (MELD scores: 11-20) and severe AH (MELD scores: 21-28).
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F-652 (Experimental): Participants will receive 10 μg/kg, 30 μg/kg or 45 μg/kg of F-652 on Day 1 and Day 7 via slow intravenous infusion. Three patients with MELD 11-20 will receive 10 μg/kg of F-652. Pharmacokinetic testing will be completed on these subjects. If evaluations demonstrate safety and efficacy signals, the next 3 patients will receive 30 μg/kg. If pharmacokinetic testing demonstrates safety and efficacy signals, the next 3 patients will receive 45 μg/kg. After demonstrating absence of side effects in this group, patients in MELD 21-28 will follow the same dose escalation regiment as the MELD 11-20 group.
  Interventions: Drug: F-652

INTERVENTIONS:
Drug: F-652 — Participants will receive 10 μg/kg, 30 μg/kg or 45 μg/kg of F-652 on Day 1 and Day 7 via slow intravenous infusion. Three patients will receive 10 μg/kg of F-652. Pharmacokinetic testing will be completed on these subjects. If evaluations demonstrate safety and efficacy signals, the next 3 patients will receive 30 μg/kg. If pharmacokinetic testing demonstrates safety and efficacy signals, the next 3 patients will receive 45 μg/kg.

SUMMARY:
Alcoholic hepatitis is a syndrome of progressive inflammatory liver injury associated with long-term heavy intake of ethanol. The pathogenesis is not completely understood. Patients who are severely affected present with subacute onset of fever, hepatomegaly, leukocytosis, marked impairment of liver function (e.g., jaundice, coagulopathy), and manifestations of portal hypertension (e.g., ascites, hepatic encephalopathy, variceal hemorrhage). However, milder forms of alcoholic hepatitis often do not cause any symptoms.

Alcoholic hepatitis usually persists and progresses to cirrhosis if heavy alcohol use continues. If alcohol use ceases, alcoholic hepatitis resolves slowly over weeks to months, sometimes without permanent sequelae but often with residual cirrhosis.

F-652 is a recombinant fusion protein containing human interleukin 22 (IL-22) and human Immunoglobulin G2 (IgG2)-Fc produced in CHO cells in serum-free culture. F-652 under development is intended to treat patients with graft vs host disease (GvHD) after bone marrow transplantation, and acute alcoholic hepatitis (AAH), a severe form of alcoholic liver disease (ALD). Both GvHD and AAH are diseases with unmet medical need. The current investigational new drug (IND) application is to conduct a phase Ia clinical study in GvHD patients to evaluate the safety and pharmacokinetic profile, and biomarkers of F-652 treatment by intravenous infusion (IV).

IL-22 is a member of the IL-10 family of cytokines which control bacterial infection, homeostasis, and tissue repair. IL-22 may be used to treat patients with ALD because of its antioxidant, anti-apoptotic, anti-steatotic, anti-microbial, and proliferative effect that have been demonstrated in various experimental systems.

DETAILED DESCRIPTION:
IL-22 is a member of the IL-10 family of cytokines which control bacterial infection, homeostasis, and tissue repair. IL-22 may be used to treat patients with ALD because of its antioxidant, anti-apoptotic, anti-steatotic, anti-microbial, and proliferative effect that have been demonstrated in various experimental systems.

The sponsor has developed F-652, a recombinant human IL-22 IgG2 Fc fusion protein produced in serum-free culture of Chinese Hamster Ovary (CHO) cells. F-652 is able to protect tissue from damage and enhance tissue repair during the inflammation process and infection by activation of STAT3 mediated by the interleukin-22 receptor subunit 1 (IL-22R1) expressed on epithelial cells such as hepatocytes.

ELIGIBILITY:
3.1 Inclusion Criteria

To participate in this study, patients must meet all of the following criteria:

1. Able to provide written informed consent (either from patient or patient's legally acceptable representative)
2. Male or female patients 21 years of age or older
3. Patients with alcoholic hepatitis defined as:

   1. History of heavy alcohol abuse use: >40 g/day in females and >60 g/day in males for a minimum period of 6 months
   2. Consumed alcohol within 6 weeks of entry into the study
   3. Serum bilirubin > 3mg/dL AND AST >ALT, but less than 500 U/L
   4. MELD score between 11-28
   5. Liver biopsy will be carried out to confirm diagnosis in all patients except those who meet criteria a-c and in whom other causes of liver disease have been excluded (viral, drug, autoimmune etc).
4. Women of child-bearing potential must utilize appropriate birth control. *Patients on steroids and/or pentoxifylline will not be excluded from the study.

Exclusion Criteria

1. Other or concomitant cause of liver disease as a result of:

   1. Autoimmune liver disease
   2. Wilson disease
   3. Vascular liver disease
   4. Drug induced liver disease Note: Concurrent viral hepatitis is not excluded.
2. Co-infection with human immunodeficiency virus (HIV)
3. Any active malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas) or any other malignancy diagnosed within the last five years.
4. Active tuberculosis on chest x-ray at study entry
5. Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, serious psychiatric disease, that, in the opinion of the Investigator would preclude the patient from participating in and completing the study
6. Patients requiring the use of vasopressors or inotropic support
7. Liver biopsy, if carried out, showing findings not compatible with alcoholic hepatitis
8. Any patient that has received any investigational drug or device within 30 days of dosing or who is scheduled to receive another investigational drug or device in the course of the study Note: Investigational drug includes any drug that is used off-label.
9. If female, known pregnancy, or has a positive urine or serum pregnancy test, or lactating/breastfeeding
10. Serum creatinine >2.5 mg/dL

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Shah, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hassanein T, McClain CJ, Vatsalya V, Stein LL, Flamm SL, Martin P, Cave MC, Mitchell M Jr, Barton B, Nagy L, Szabo G, McCullough A, Dasarathy S, Shah J, Blevins C, Scott D, Krebs W, Brown JE, Lin W. Safety, Pharmacokinetics, and Efficacy Signals of Larsucosterol (DUR-928) in Alcohol-Associated Hepatitis. Am J Gastroenterol. 2024 Jan 1;119(1):107-115. doi: 10.14309/ajg.0000000000002275. Epub 2023 Apr 3. PMID 37011138

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: F-652 10 μg/kg: Participants will receive 10 μg/kg of F-652 on Day 1 and Day 7 via slow intravenous infusion.
- Period 2: F-652 30 μg/kg: Participants will receive 30 μg/kg of F-652 on Day 1 and Day 7 via slow intravenous infusion.
- Period 3: F-652 45 μg/kg: Participants will receive 45 μg/kg of F-652 on Day 1 and Day 7 via slow intravenous infusion.
Period: Overall Study
Arm/Group | Period 1: F-652 10 μg/kg | Period 2: F-652 30 μg/kg | Period 3: F-652 45 μg/kg
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: F-652 10 μg/kg | Period 2: F-652 30 μg/kg | Period 3: F-652 45 μg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (6.9) | 50.5 (12.0) | 50.3 (11.3) | 49.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 4 | 4 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 6 | 6 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18
Alcohol Consumption by MELD grouping [Mean (Standard Deviation); unit: grams per day] — Amount of alcohol consumed on a daily basis measured in grams. A MELD score (model for end state liver disease) ranks the degree of sickness the degree to which a liver transplant is needed. The higher the number the more severe the sickness and the more urgent need for a liver transplant. Population: The six participants in each period were further defined by MELD grouping, where three participants had a MELD score of 11-20 and three participants had a MELD score of 21-28; resulting in a total of six participants in each period, a total of 18 subjects overall.
  grams per day
    MELD 11-20: number analyzed (Participants) | 3 | 3 | 3 | 9
    MELD 11-20 | 143.3 (75.0) | 151.3 (28.8) | 186.6 (88.9) | 160.4 (63.1)
    MELD 21-28: number analyzed (Participants) | 3 | 3 | 3 | 9
    MELD 21-28 | 181.3 (140.0) | 212.6 (141.7) | 57.3 (28.0) | 150.4 (123.2)
Hospitalized at screening by MELD grouping [Count of Participants; unit: Participants] — Number of subjects hospitalized at screening visit. A MELD score (model for end state liver disease) ranks the degree of sickness the degree to which a liver transplant is needed. The higher the number the more severe the sickness and the more urgent need for a liver transplant. Population: The six participants in each period were further defined by MELD grouping, where three participants had a MELD score of 11-20 and three participants had a MELD score of 21-28; resulting in a total of six participants in each period, a total of 18 subjects overall.
  Participants
    MELD 11-20: number analyzed (Participants) | 3 | 3 | 3 | 9
    MELD 11-20 | 3 | 3 | 2 | 8
    MELD 21-28: number analyzed (Participants) | 3 | 3 | 3 | 9
    MELD 21-28 | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Unexpected Serious Adverse Events.
Description: The count of subjects who experience serious adverse events
Time Frame: From day 1 up to 42 days following administration of last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: F-652 10 μg/kg | Period 2: F-652 30 μg/kg | Period 3: F-652 45 μg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 42 days following the last administration of study treatment for each subject, an average of 56 days
Arm/Group | Period 1: F-652 10 μg/kg | Period 2: F-652 30 μg/kg | Period 3: F-652 45 μg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 5/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: F-652 10 μg/kg (N=6) | Period 2: F-652 30 μg/kg (N=6) | Period 3: F-652 45 μg/kg (N=6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Leukocytosis (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tremors (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Weakness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Increased body temperature (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT02655510/Prot_SAP_000.pdf